CLINICAL TRIAL: NCT07334223
Title: Comparison of Intravenous Ondansetron and Low Dose Ketamine in Preventing Post Spinal Shivering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Hospital Lahore (Other)
Responsible Party: Principal Investigator, Adeel Ahmed, Principal Investigator, Mayo Hospital Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mayo1
Record Dates: First submitted 2026-01-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Shivering; Postspinal Shivering
Keywords: Spinal anesthesia; Postoperative shivering; Shivering prophylaxis; Ondansetron; Ketamine
MeSH Terms: interventions — Ondansetron; Ketamine; N-methyl-d-aspartate receptor antagonist MN-08

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Ondansetron (Experimental): Received 8 mg of ondansetron administered intravenously five minutes after spinal anesthesia for prophylaxis of post spinal shivering.
  Interventions: Drug: ondansetron
- Group Low Dose Ketamine (Active Comparator): Received ketamine 0.25 mg per kilogram administered intravenously five minutes after spinal anesthesia for prophylaxis of post spinal shivering.
  Interventions: Drug: Ketamine (0.25 mg/kg)

INTERVENTIONS:
Drug: ondansetron — 8 mg ondansetron administered intravenously as a single dose five minutes after spinal anesthesia.
  Other Names: Serotonin type 3 receptor antagonist
  Arms: Group Ondansetron
Drug: Ketamine (0.25 mg/kg) — 0.25 mg per kilogram ketamine administered intravenously as a single dose five minutes after spinal anesthesia.
  Other Names: N-methyl-D-aspartate receptor antagonist
  Arms: Group Low Dose Ketamine

SUMMARY:
This randomized controlled trial assessed whether intravenous ondansetron is more effective than low dose ketamine in preventing shivering after spinal anesthesia in adults undergoing elective surgery. Post spinal shivering is a frequent and uncomfortable complication of spinal anesthesia and may increase oxygen demand and interfere with routine monitoring. Adults aged 20 to 70 years (body weight 50 to 80 kg; American Society of Anesthesiologists class I to II) scheduled for elective procedures under standardized spinal anesthesia were randomly allocated in equal numbers to receive either ondansetron 8 mg intravenously or ketamine 0.25 mg/kg intravenously, administered 5 minutes after the spinal injection. Perioperative temperature management was standardized for all participants. The primary outcome was the occurrence of post spinal shivering during intraoperative monitoring. Among 180 participants, shivering occurred in 30.0% of those receiving ondansetron and 44.4% of those receiving ketamine, showing a statistically significant reduction with ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender aged 20-60 years with ideal body
* weight of 50 to 80 kg.
* Patients meeting ASA classification I and II determined by
* anesthesiologist.
* Patients undergoing elective surgeries under spinal anesthesia.
* Duration of surgery should not be more than 3 hours.

Exclusion Criteria:

* Patients having a documented history of severe adverse reactions to ketamine or ondansetron.
* Patients with cardiovascular disease documented in history.
* Patients with hepatic disease documented in history and supported by lab results (AST 32-40U/L), ALT(10-40U/L).
* Patients with renal disease documented in history and supported by lab results. Urea (10-50mg/dl) S/Creatinine (0.3-1.5mg/dl).
* Patients with hyperthyroidism documented in history and supported by lab results.
* Patients with history of mental illness, seizures and glaucoma.
* Patients with known hypertension (BP greater than 140/90).
* Haemodynamically unstable patients (BP<100mmHg).
* Patients with coagulopathy or other bleeding diathesis documented in history and supported by lab results.
* Complicated prolonged surgeries in spinal anesthesia.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency of Post Spinal Shivering | From 5 minutes after administration of study drug until transfer of the patient to the post-anesthesia care unit
  Occurrence of post spinal shivering following administration of study medication, assessed clinically by the anesthesiology team and recorded as present or absent during intraoperative monitoring after spinal anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Ahmed, Principal Investigator — Mayo Hospital Lahore
Locations (1):
- Mayo Hospital, Lahore, Lahore, Punjab Province, Pakistan